CLINICAL TRIAL: NCT02137811
Title: Chart Review of Demographics and Clinical Outcomes and Physician Attitudes in Patients Who Have Received the Microculture Kinetic (MiCK) Apoptosis Test
Brief Title: Demographics, Clinical Outcomes, and Physician Attitudes in Patients Who Have Received The MiCK Assay (CorrectChemo)
Status: Withdrawn | Type: Observational
Why Stopped: Company decided to remove CLIA test from Market.
Sponsor: Pierian Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 1143088; 187128 (Other Grant/Funding Number: DiaTech)
Record Dates: First submitted 2014-04-23; First posted 2014-05-14 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
Keywords: cancer; CorrectChemo; assay; lab test; MICK assay; apoptosis; increase survival; increase response rates; decrease time to progression; chemotherapy; cancer treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients that received MICK assay: Patients with pathological diagnoses of cancer or leukemia who have had a MiCK assay (CorrectChemo) test performed
  Interventions: Other: MICK Assay

INTERVENTIONS:
Other: MICK Assay — An automated microculture kinetic (MiCK) assay for measuring drug induced apoptosis in tumor cells; the MiCK assay for apoptosis provides a mechanism-based approach to studying effects of cytotoxic agents on tumor cells.
  Other Names: CorrectChemo

SUMMARY:
Recently an automated test for measuring cancer cell death in the presence of chemotherapy has been developed. This test has been called the MiCK assay during the ten year development phase and is now called Correct Chemo.

CorrectChemo provides the medical community and patients a way to determine the effects of different chemotherapies on individual cancer cells.

MiCK assay has been proven to have clinical usefulness in two studies. In one study using multiple types of cancer, physicians used the MiCK assay in 63% of the patients. If the physician used the results to prescribe the chemotherapy treatment, the patients' response rate, time to the disease getting worse, and overall survival were all significantly better compared to patients whose physicians did not use the results. In another study of breast cancer patients, physicians used the MiCK assay in 74% of patients. If the results were used when planning chemotherapy, response rate and time to the disease started getting worse were all significantly better compared to patients whose physicians did not use the results of the MiCK assay The purpose of this study is to compare the outcomes of patients who have had the MiCK assay (CorrectChemo) with tumor types, physician attitudes towards the test, and how the physicians used the test. This study will be gathering this data by reviewing medical charts.

DETAILED DESCRIPTION:
The purpose of this study is to correlate the clinical outcomes of patients who have had the MICK assay with tumor type, physician attitudes towards the assay, and how physicians used the assay by using data in patient charts, and surveying physician attitudes.

Study Objectives:

1. To determine how often physicians use the MiCK assay results in developing a treatment plan, and which drugs the physician used in treatment. This will be correlated with patient and tumor demographics.
2. To determine physician attitudes towards the MiCK assay.
3. To determine the clinical outcomes (response rates, time to progression, and overall survival) in patients who have had a MiCK assay. This will be correlated with pattern of physician use of the assay.

Treatment Plan:

1. The treating oncologist will provide demographic information (patient identifying number, sex, age, number of prior lines of therapy, performance status) and tumor information (cell type, stage, metastatic sites, goal of therapy, pre-assay planned therapy, and post-assay therapy chosen for
2. Tumor response, patient symptom response, time to progression on each chemotherapy regimen, and overall survival will be determined from the patient chart and will be correlated with MICK assay results.
3. Physicians will complete a questionnaire on attitudes towards usefulness of the assay.

Statistics

1. Investigators will correlate tumor response, symptom response, time to progression and overall survival with drug therapy with drug response in MICK assay for first chemo regimen after assay, and according to pattern of physician use of the assay.
2. We will accumulate physician attitudes toward usefulness of the assay.

Informed Consent Since this study has no risk to the patient, informed consent will not be needed. Physicians will have the option of participating, or not participating, in each patient. Physicians will be compensated for completing chart review and submitting data after the MiCK assay has been performed, and at 6,12 and 24 months after MiCK assay.

Data Collection from Physicians Data will include demographics and tumor characteristics and physician attitudes: I used the test to develop a treatment plan yes/no, I found the test useful yes/no, I found the test to be helpful in planning for palliative care yes/no, I found the test to be helpful in planning for hospice yes/no. I have these suggestions for improvement (free text response). Data will include at 6,12 and 24 months clinical outcomes as judged by the physician: Complete, Partial, Stable, Death, symptomatic improvement patient felt better same or worse. Data will include at time of progression, did doctor use the MiCK assay to plan the next treatment, try to get another MiCK assay, or use the assay to plan for palliative care or hospice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological diagnoses of cancer or leukemia who have had a MiCK assay (Correct Chemo) performed

Exclusion Criteria:

* Patients whose physician refuses to provide data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathological diagnoses of cancer or leukemia who have had a MiCK assay (CorrectChemo) performed
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Clinical composite outcomes | 6 months
  To determine the clinical outcomes (response rates, time to progression, and overall survival) in patients who have had a MiCK assay (CorrectChemo.) This will be correlated with pattern of physician use of the assay.
Clinical composite outcomes | 12 months
  To determine the clinical outcomes (response rates, time to progression, and overall survival) in patients who have had a MiCK assay (CorrectChemo). This will be correlated with pattern of physician use of the assay.
Clinical composite outcomes | 24 months
  To determine the clinical outcomes (response rates, time to progression, and overall survival) in patients who have had a MiCK assay (CorrectChemo.) This will be correlated with pattern of physician use of the assay.

SECONDARY OUTCOMES:
How often Physicians use MiCK assay (CorrectChemo) results in patient treatment plan | 6 months
  To determine how often physicians use the MiCK assay (CorrectChemo) results in developing a treatment plan, and which drugs the physician used in treatment. This will be correlated with patient and tumor demographics.
How often Physicians use MiCK assay (CorrectChemo) results in patient treatment plan | 12 months
  To determine how often physicians use the MiCK assay (CorrectChemo) results in developing a treatment plan, and which drugs the physician used in treatment. This will be correlated with patient and tumor demographics.
How often Physicians use MiCK assay (CorrectChemo) results in patient treatment plan | 24 months
  To determine how often physicians use the MiCK assay (CorrectChemo) results in developing a treatment plan, and which drugs the physician used in treatment. This will be correlated with patient and tumor demographics.

OTHER OUTCOMES:
Physician attitudes | 6 months
  To determine how often physicians use the MiCK assay (CorrectChemo)results in developing a treatment plan, and which drugs the physician used in treatment. This will be correlated with patient and tumor demographics.
Physician attitudes | 12 months
  To determine how often physicians use the MiCK assay (CorrectChemo)results in developing a treatment plan, and which drugs the physician used in treatment. This will be correlated with patient and tumor demographics.
Physician attitudes | 24 months
  To determine how often physicians use the MiCK assay (CorrectChemo)results in developing a treatment plan, and which drugs the physician used in treatment. This will be correlated with patient and tumor demographics.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Hallquist, MD, Principal Investigator — Pierian Biosciences
Locations (2):
- DiaTech Oncology, Franklin, Tennessee, United States
- DiaTech Oncology, Montreal, Quebec, Canada